CLINICAL TRIAL: NCT00405392
Title: An Open-label, Multi-centre, Randomized Study to Investigate Patient Preference on Dosing in the Once-monthly Ibandronate and the Once-weekly Risedronate in Korean Women With Postmenopausal Osteoporosis. A Six-month, Two-sequence, and Two Period Crossover Study
Brief Title: Study To Investigate Patient Preference On Dosing In Ibandronate And Risedronate In Korean Women With Postmenopausal Osteoporosis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 109393
Record Dates: First submitted 2006-11-29; First posted 2006-11-30 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-03

CONDITIONS: Osteoporosis, Postmenopausal
Keywords: risedronate; Ibandronate; preference; Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — Ibandronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Ibandronate (SB743830HD)

SUMMARY:
This is a randomized open label, multi-centre study for Korean women with postmenopausal osteoporosis, evaluating the preference for either the once-monthly dosing of ibandronate or the once-weekly dosing of risedronate.

Eligible subjects will be randomised either ibandronate monthly regimen or risedronate weekly regimen.

Treatment period consists of 3 month with ibandronate 150mg and additional 12 week with risedronate 35 mg or vice versa.

After taking the first interventional medicine for 3 months or 12 weeks completely, a subject changes the treatment arm. There is no washout period.

ELIGIBILITY:
Inclusion Criteria:

* Women with postmenopausal osteoporosis diagnosed by DXA scanning, defined by T-score of -2.5 SD at spine or femur.
* Patients who have never received bisphosphonates therapy (bisphosphonates naive)

Exclusion Criteria:

* Inability to stand or sit in the upright position for at least 60 minutes;
* Hypersensitivity to any component of risedronate and ibandronate;
* Administration of any investigational drug within 30 days preceding the first dose of the study drug;
* Patient has been on hormone (estrogen) replacement therapy or other osteoporosis medication (e.g. SERMS and calcitonin) within the previous 3 months.
* Patient has been on systemic corticosteroids therapy for more than 1 month within the past year.
* Other bone disease except osteoporosis
* Current medical history of uncontrolled major upper GI disease

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2007-03-22 (Actual); Primary Completion 2008-05-27 (Actual); Study Completion 2008-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 365 korean female participants with postmenopausal osteoporosis were enrolled in this study, conducted for 6 months at 15 centers in South Korea.
Pre-assignment Details: A total of 365 participants were randomized in the study. Out of the randomized participants 13 were dropped out before administration of drug, remaining 352 participants were included in safety population, 314 participants were included in modified intent to treat population and 308 participants were included in the per-protocol population.
Groups:
- Sequence A: Ibandronate 150 mg Then Risedronate 35 mg: Participants received treatment of ibandronate 150 milligram (mg) tablet orally once monthly for 3 months in period 1 and then administered risedronate 35 mg tablet orally once weekly for 12 weeks in period 2 in sequence A. Participants were recommended to take the tablet on the same day every month in case of the once-monthly drug (e.g. on the 15th each month) and on the same day every week in case of the once-weekly drug (e.g. every Sunday). The two drugs were administered on an empty stomach in the morning, followed by an overnight fast (at least 6-hour fast).
- Sequence B: Risedronate 35 mg Then Ibandronate 150 mg: Participants received treatments of risedronate 35 mg tablet orally once weekly for 12 weeks in period 1 and then administered ibandronate 150 mg tablet orally once monthly for 3 months in period 2 in sequence B. Participants were recommended to take the tablet on the same day every month in case of the once-monthly drug (e.g. on the 15th each month) and on the same day every week in case of the once-weekly drug (e.g. every Sunday). The two drugs were administered on an empty stomach in the morning, followed by an overnight fast (at least 6-hour fast).
Period: Overall Study
Arm/Group | Sequence A: Ibandronate 150 mg Then Risedronate 35 mg | Sequence B: Risedronate 35 mg Then Ibandronate 150 mg
Started | 183 | 182
Completed | 153 | 155
Not Completed | 30 | 27
Not completed — Adverse Event | 15 | 14
Not completed — Did not meet Eligibility criteria | 7 | 2
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Data missing | 2 | 0
Not completed — Non-compliance | 0 | 1
Not completed — Other | 1 | 5

BASELINE CHARACTERISTICS:
Population: Safety population: Any participant who was administered with the study drug once more and had safety information was included in the safety analysis population regardless of early termination.
Groups:
- Sequence A: Ibandronate 150 mg Then Risedronate 35 mg: Participants received treatment of ibandronate 150 mg tablet orally once monthly for 3 months in period 1 and then administered risedronate 35 mg tablet orally once weekly for 12 weeks in period 2 in sequence A. Participants were recommended to take the tablet on the same day every month in case of the once-monthly drug (e.g. on the 15th each month) and on the same day every week in case of the once-weekly drug (e.g. every Sunday). The two drugs were administered on an empty stomach in the morning, followed by an overnight fast (at least 6-hour fast).
- Total: Total of all reporting groups
Arm/Group | Sequence A: Ibandronate 150 mg Then Risedronate 35 mg | Sequence B: Risedronate 35 mg Then Ibandronate 150 mg | Total
Number analyzed (Participants) | 176 | 176 | 352
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.33 (6.53) | 61.99 (7.07) | 61.66 (6.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 176 | 176 | 352
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  South Korea | 176 | 176 | 352

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Prefer the Once-monthly Dosing of Ibandronate to the Once-weekly Dosing of Risedronate
Description: Preference of monthly ibandronate and weekly risedronate was compared. Modified-intention-to-treat (mITT) population was used for analysis. Any participant randomly assigned, received the study drug, and participants were asked to fill the preference questionnaire on completion of study. Preference was calculated as percentage. Data for percentage of participants with preference to once-monthly dosing of ibandronate to the once-weekly dosing of risedronate was presented.
Time Frame: Visit 4 (Week 24)
Population: mITT population was comprised of any participant, who was randomly assigned, received the study drug once more at each phase, filled out the preference questionnaire at the completion of the study. Percentages do not sum to 100 because some participants did not express a preference.
Measure: Number; unit: Percentage of participants
Groups:
- Ibandronate 150 mg Once Monthly: Participants received ibandronate 150 mg tablet orally once in a month for 3 months either in period 1 or period 2 as per the randomization sequence. Participants were recommended to take the tablet on the same day every month in case of the once-monthly drug (e.g. on the 15th each month). The treatment was administered on an empty stomach in the morning, followed by an overnight fast (at least 6-hour fast).
- Risedronate 35 mg Once Weekly: Participants received risedronate 35 mg tablet orally once weekly for 12 weeks either in period 1 or period 2 as per the randomization sequence. Participants were recommended to take the tablet on the same day every month in case of the once-monthly drug (e.g. on the 15th each month). The treatment was administered on an empty stomach in the morning, followed by an overnight fast (at least 6-hour fast).
Arm/Group | Ibandronate 150 mg Once Monthly | Risedronate 35 mg Once Weekly
Number analyzed (Participants) | 314 | 314
Percentage of participants | 62.42 | 21.02
Statistical Analysis 1: Comparison: Ibandronate 150 mg Once Monthly vs Risedronate 35 mg Once Weekly; Test type: Superiority or Other; p < 0.0001, Chi-squared

2. Secondary Outcome: Percentage of Participants Choosing Ibandronate or Risedronate as Their Preferred Treatment Based on Convenience of Administration
Description: Participant's preference for convenient treatment was compared between monthly ibandronate and weekly risedronate. Analysis population was mITT. Preference for convenient treatment was calculated as percentage. Percentage of participants who think once-monthly ibandronate dosing is more convenient over once-weekly risedronate dosing were presented. Those participants who answered the two treatments equally convenient were excluded while reporting.
Time Frame: Visit 4 (Week 24)
Population: mITT Population. Percentages do not sum to 100 because some participants did not express a preference.
Measure: Number; unit: Percentage of particiants
Arm/Group | Ibandronate 150 mg Once Monthly | Risedronate 35 mg Once Weekly
Number analyzed (Participants) | 314 | 314
Percentage of particiants | 72.93 | 13.69
Statistical Analysis 1: Comparison: Ibandronate 150 mg Once Monthly vs Risedronate 35 mg Once Weekly; Test type: Superiority or Other; p < 0.0001, Chi-squared

3. Secondary Outcome: Mean Percent Change of Serum C-terminal Telopeptide (CTx) From Baseline to Visit 3 for Once-monthly Dosing of Ibandronate & Once-weekly Dosing of Risedronate
Description: The difference of change in serum CTX from basal value between the two sequences was tested using ANCOVA at 95% confidence interval at 3 months (Visit 3) after the administration. Analysis was done with PP population. Baseline was value at Week 0, Change from baseline was calculated by subtracting Baseline value from value at specified time point.
Time Frame: Baseline (Week 0) and Visit 3 (Week 12)
Population: Per protocol population comprised of any participant, who didn't violate the study protocol, filled the preference questionnaire at the completion of the study, finished assessment of bone turnover marker, and completed journal of GI symptoms. Only the participants available at the time of assessment were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Ibandronate 150 mg Once Monthly | Risedronate 35 mg Once Weekly
Number analyzed (Participants) | 153 | 154
Percent change | -57.23 (35.89) | -56.95 (37.07)
Statistical Analysis 1: Comparison: Ibandronate 150 mg Once Monthly vs Risedronate 35 mg Once Weekly; Test type: Superiority or Other; p = 0.9456, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Up to 6 months
Description: Safety population was used to analyze adverse events and all-cause mortality. Datasets could not be located to generate separate non-serious adverse event table.
Arm/Group | Ibandronate 150 mg Once Monthly | Risedronate 35 mg Once Weekly
All-Cause Mortality (participants affected / at risk) | 0/336 | 0/334
Serious Adverse Events (participants affected / at risk) | 6/336 | 4/334
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibandronate 150 mg Once Monthly (N=336) | Risedronate 35 mg Once Weekly (N=334)
Intervertebral Disc Disorder (Musculoskeletal and connective tissue disorders) | 2 | 0
Varicose vein operation (Surgical and medical procedures) | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Aspergilloma (Infections and infestations) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 2
Papillary thyroid cancer (Endocrine disorders) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.